CLINICAL TRIAL: NCT05228418
Title: Bridging ED to Outpatient AUD Therapy With Naltrexone
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Principal Investigator, David Hui, Resident Physician, Albert Einstein Healthcare Network
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-546
Record Dates: First submitted 2022-01-14; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participant (Experimental): All participants who meet inclusion criteria will be offered oral naltrexone in the ED, a bridge prescription for oral naltrexone, and be referred to outpatient MAT clinic where participants will be offered monthly IM naltrexone injections.
  Interventions: Drug: Naltrexone Pill

INTERVENTIONS:
Drug: Naltrexone Pill — Naltrexone oral bridge to IM naltrexone maintenance therapy
  Other Names: naltrexone IM 380mg

SUMMARY:
Alcohol use disorder (AUD) is a treatable and common condition encountered in the emergency department, but unfortunately is rarely directly addressed in emergency departments nationwide. To our knowledge, initiation of medication assisted therapy (MAT) for AUD in the emergency department setting has not been widely adopted. Our project is novel for its scope to use a medication well-tested in the outpatient environment and bring it to the emergency department in order to more effectively link patients to outpatient alcohol use reduction therapy as part of a medication assisted therapy (MAT). The investigators are proposing a feasibility project to initiate oral naltrexone to eligible ED patients deemed to have alcohol use disorder and who are interested in cutting down their drinking. The investigators plan to connect these patients with outpatient follow-up in our own community practice center (CPC) for intramuscular (IM) Vivitrol injections under the supervision of the Einstein Toxicology Department. Through the CPC, patients can also be referred to other supporting services such as Alcoholics Anonymous for multidisciplinary care. The investigators are optimistic that this innovative warm hand off from the initial ED visit to outpatient follow-up will ultimately decrease problematic drinking, improve patient's health, and benefit the hospital.

Our main objective is to establish a pathway to encourage patients who present to the emergency room with acute sequelae of alcohol use disorder to enter outpatient treatment. Our intervention will be the initiation of oral naltrexone with warm handoff to the Community Practice Center where patients will be transitioned to intramuscular (IM) Vivitrol for chronic maintenance therapy. Thus success will be measured by primarily: percentage of patients who make it to their first outpatient visit for the Vivitrol injection, percentage of patients who continue with treatment and continue to receive Vivitrol for their second injection.

DETAILED DESCRIPTION:
The burden of excessive alcohol use in Pennsylvania is significant. In 2013, the CDC estimated that excessive alcohol use caused about 3,510 deaths per year in Pennsylvania and cost an estimated $8.3 billion annually, or $1.81 per alcoholic drink consumed. An internal query of the Einstein Medical Center Philadelphia emergency department database found that, during a 12-month period spanning 2019-2020, 1,568 patients were discharged with an ICD-10 diagnosis related to alcohol use. This equates to approximately 1.6% of all Einstein Philadelphia emergency department ED visits being directly related to alcohol use. Currently, there is no standard of care for treatment of alcohol use disorder in the emergency department. To address this community need for an ED based intervention, the investigators propose the administration of Vivitrol, which is a medication that has been shown to reduce heavy alcohol drinking by as much as 25% compared to placebo in one study by Garbutt et al. Bryson et al found that patients who received Vivitrol injections were more likely to continue with treatment and decrease non-pharmacological healthcare costs, including inpatient hospitalizations and emergency department visits. This intervention has already been successfully implemented in at least one hospital in California as reported by Anderson et al. Vivitrol assisted warm hand-off to outpatient medication assisted therapy (MAT) may be an evidence-based approach to give this high-risk ED patient population a reliable mechanism to reduce their problematic drinking. This will benefit both public health and alleviate the burden of alcohol use in our ED.

Patients will be recruited from the Emergency Department of Einstein Medical Center Philadelphia. The Einstein Medical Center Philadelphia is an urban teaching hospital, level one trauma center with 500 beds and an annual emergency department census of 98,000 subjects. Patients will be asked to follow-up in the medication assisted treatment (MAT) clinic located in the community practice clinic (CPC), which is also located at Einstein Medical Center Philadelphia. Those interested in reducing or stopping their alcohol use are potential subjects in this study. The Division of Clinical Research of the Department of Emergency Medicine has extensive experience in both investigator led and pharmaceutical research. Einstein Medical Center emergency department has research associates on site five days a week who will perform the retrospective study and enroll eligible subjects.

This is primarily a study to evaluate the feasibility of a novel process to screen, educate, and initiate oral naltrexone for treatment of patients with alcohol use disorder who are interested in the reduction or complete cessation of their drinking. The ultimate goal is to transition patients to long term outpatient treatment with intramuscular naltrexone. Potential patients will be identified by the ED clinical care team. In-house research associates will screen for inclusion and exclusion criteria, and they will also consent the patients. Patients will have blood drawn for hepatic function test studies and urine collected for urine drug screen with expanded opioid panel as part of the drug manufacturer's recommended protocol. Patients who are enrolled in the study will complete a short intake survey, be given their first dose of naltrexone in the ED, and be discharged with a week's prescription for a daily 50mg dose of oral naltrexone, which is the standard dose for treatment of alcohol use disorder. Patients will also receive a follow-up appointment in the MAT (medication assisted therapy) clinic located in the CPC within 1 week of the index ED visit. Patients will be prescribed IM naltrexone 380mg (Vivitrol) which will be administered that visit and any subsequent monthly follow-up visits. Patients will be called on their cell phone with a reminder prior to the clinic visit.

The research associates as well as the health care team (both residents and attending physicians) will screen patients who present to the ED with any complaint that could be related to alcohol use disorder. These patients may be initially intoxicated. Once patients are judged to be clinically sober by the emergency department team, they will be assessed for whether they are interested in reducing their alcohol use through pharmacological intervention and warm hand off to Einstein's outpatient MAT clinic. Patients who are interested in enrolling in this study will be assessed for appropriateness by the research team during normal weekday business hours. An important aspect of the inclusion criteria will be to screen for problematic drinking based on the AUDIT score, which is an international used 10 item survey used to risk stratify patients for harmful alcohol use. A score of 16 or higher suggests high risk for problematic alcohol use. An AUDIT score greater than this threshold in combination with a patient who has already experienced a consequence of drinking to the point that he or she has presented to the emergency room strongly suggests to us that the patient may benefit from rapid outpatient follow-up and be started on medication assisted treatment. After training, the emergency department licensed social worker and/or certified recovery specialist may assist the research associate in screening and assessing these patients.

A standardized data collection form will be used to collect intake clinical data. Initial data gathered will include age, gender (male, female, other), race/ethnicity (White, American Indian and Alaska Native, Asian, Black or African American, Native Hawaiian and other Pacific Islander, other), current employment (yes/no), highest level of education (high school, bachelors, masters, phd/equivalent, other). Data obtained in follow-up clinic visits will be entered into the patient's medical chart to be used as part of their usual clinical care for management of their alcohol use disorder. This data will be abstracted by research associates in a deidentified manner. The investigators will also track the total cost of IM naltrexone not covered by the patient's insurance. Data will be stored for 6 years after the completion of the study.

A pre-intervention survey will be administered at the index emergency department visit after patients are enrolled successfully into the study, and follow-up survey will be administered in the clinic as part of a semi-standardized initial clinic visit and the follow-up clinic visit four-weeks later. Patients' drinking behaviors and alcohol cravings will be assessed based on a questionnaire adapted from externally validated surveys, such as the Penn Alcohol Craving Scale. Success will be judged based on how many patients ultimately follow-up through our proposed naltrexone assisted warm handoff process. The primary endpoint is percentage of patients who are successfully referred to outpatient MAT treatment in our CPC clinic and percentage of people who stay in treatment at the follow-up outpatient clinic visit. Other secondary includes tracking variables that the investigators believe to correlate with alcohol use disorder, such as estimation of alcohol intake, cravings, based on standardized surveys administered during the MAT clinic visits. Additionally, the investigators will be collecting a whole host of demographic and substance use history to see if there are any factors that are associated with failure to retain patients in treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Presents to the ED with chief complaint of alcohol use or judged to have alcohol use as a significant contributing factor to their presentation to the emergency department
* Patients must be interested in reducing or stopping their alcohol use
* AUDIT score greater or equal to 16

Exclusion Criteria:

* Patients will be excluded if they previously participated in the study
* patients who will be admitted to the hospital
* Endorse dependence on opioid medications or opioid street drugs
* have an extended urine drug screen that is positive for opioids
* elevated liver transaminase (AST or ALT) that is greater than 5 times the upper limit of normal
* decompensated liver disease
* allergic reaction to naltrexone
* pregnant
* prisoners
* unable to provide consent
* subjects in police custody
* non-English speaking
* have no reliable means for future contact.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Successful referral and follow-up in MAT clinic | 4 weeks
  The primary endpoint is percentage of patients who are successfully referred to outpatient MAT treatment in our hospital's outpatient clinic and percentage of people who stay in treatment at the intake and subsequent follow-up outpatient clinic visit. (i.e. % of patients who remain in treatment at the initial outpatient intake visit scheduled within 1 week of the initial index ED visit and the follow-up appointment 4 weeks after the intake visit)

SECONDARY OUTCOMES:
Alcohol use severity measures | 4 weeks
  We will track variables that we believe to correlate with alcohol use disorder, such as estimation of weekly alcohol intake, alcohol cravings cravings, ED visits for alcohol use for the previous week via surveys administered during the intake outpatient MAT visit and the follow-up appointment 4 weeks later.

CONTACTS AND LOCATIONS:
Overall Officials: David Hui, MD, Principal Investigator — Albert Einstein Medical Center
Locations (1):
- Albert Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garbutt JC, Kranzler HR, O'Malley SS, Gastfriend DR, Pettinati HM, Silverman BL, Loewy JW, Ehrich EW; Vivitrex Study Group. Efficacy and tolerability of long-acting injectable naltrexone for alcohol dependence: a randomized controlled trial. JAMA. 2005 Apr 6;293(13):1617-25. doi: 10.1001/jama.293.13.1617. PMID 15811981
- [Background] Anderson ES, Chamberlin M, Zuluaga M, Ullal M, Hawk K, McCormack R, D'Onofrio G, Herring AA. Implementation of Oral and Extended-Release Naltrexone for the Treatment of Emergency Department Patients With Moderate to Severe Alcohol Use Disorder: Feasibility and Initial Outcomes. Ann Emerg Med. 2021 Dec;78(6):752-758. doi: 10.1016/j.annemergmed.2021.05.013. Epub 2021 Aug 2. PMID 34353648
- [Background] Bryson WC, McConnell J, Korthuis PT, McCarty D. Extended-release naltrexone for alcohol dependence: persistence and healthcare costs and utilization. Am J Manag Care. 2011 Jun;17 Suppl 8(Suppl 8):S222-34. PMID 21761949